CLINICAL TRIAL: NCT01416675
Title: Delirium Assessment in the Pediatric Intensive Care Unit
Acronym: DIPI-ICU
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charite University, Berlin, Charite University, Berlin, Germany
Other Study IDs: DIPI-ICU
Record Dates: First submitted 2011-08-12; First posted 2011-08-15 (Estimated); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Pediatric Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Objective: Studies documenting the prevalence of delirium among critically ill children are still rare. Emerging literature from psychiatric specialists reports the prevalence of delirium to be approximately 10% in the pediatric intensive care unit (PICU). This is likely to be an underestimation of the true prevalence, as demonstrated in early adult delirium literature, especially given the absence of validated bedside tools to diagnose delirium in the PICU.

The primary aim of this study is to validate the German version of the Pediatric Confusion Assessment Method for the Intensive Care Unit (pCAM-ICU). The secondary aim of the study is to compare validity and reliability of the pCAM-ICU and the Pediatric Anesthesia Emergence Delirium (PAED) Scale.

ELIGIBILITY:
Inclusion Criteria:

* pediatric ICU patients

Exclusion Criteria:

* non-German-speaking
* inability to communicate due to severe hearing loss or brain injury
* preexisting psychosis
* mental retardation due to a specific diseases (e.g. M. Crouzon, Kabuki Syndrome, Z.n. Battered Child, Atrogryposes multiplex congenita)

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric Intensive Care Unit Patients
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the pediatric confusing assessment method for the intensive care unit (pCAM-ICU) | The participants will be followed up in the sample period (1 to 21 days)

SECONDARY OUTCOMES:
Specifity of the pediatric confusing assessment method for the intensive care unit (pCAM-ICU) | The participants will be followed up in the sample period (1 to 21 days)
Specifity of the Delirium Rating Scale (DRS) | The participants will be followed up in the sample period (1 to 21 days)
Sensitivity of the Delirium Rating Scale (DRS) | The participants will be followed up in the sample period (1 to 21 days)
Positive predictive value of the Delirium Rating Scale (DRS) | The participants will be followed up in the sample period (1 to 21 days)
Prevalence of delirium | The participants will be followed up in the sample period (1 to 21 days)
  Measured with pediatric confusing assessment method for the intensive care unit (pCAM-ICU), Delirium Rating Scale (DRS) and DSM-IV-criteria
Depth of sedation | The participants will be followed up in the sample period (1 to 21 days)
  Measured with Richmond Agitation Sedation Scale (RASS)
Quality of Analgesia | The participants will be followed up in the sample period (1 to 21 days)
  Measured by Face Pain Scale, Revised (FPS-R) und the Numeric Analog Scale (NAS) or COMFORT Behavior-Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, Campus Virchow Klinikum and Campus Charité mitte, Charité - Universitaetsmedizin Berlin, Berlin, Germany